CLINICAL TRIAL: NCT00224315
Title: Clozapine-Augmentation With Ziprasidone or Risperidone, a Randomized, Prospective Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZR-zink
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Schizophrenia, Schizoaffective Disorder
Keywords: Schizophrenia,; schizoaffective disorder,; treatment resistancy; clozapine,; ziprasidone; risperidone; combination
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — ziprasidone; Risperidone

INTERVENTIONS:
Drug: ziprasidone
Drug: risperidone

SUMMARY:
We aim to compare the augmentation of clozapine with ziprasidone or risperidone in a randomized, prospective manner.

DETAILED DESCRIPTION:
Partial response of schizophrenic psychoses to a monotherapy with clozapine is a frequent problem of clinical psychiatry. Current problems are treatment resistant positive and/or negative symptoms, as well as side effects. Therefore, different strategies of augmentations have been applied. Based on successful experiences in case reports and results of other work groups, we aim to compare the augmentation of clozapine with ziprasidone or risperidone in a randomized, prospective manner.

ELIGIBILITY:
Inclusion Criteria:

* Treatment resistant schizophrenic or schizoaffective disorder under therapy with clozapine,
* Age between 18 and 70,
* Informed consent

Exclusion Criteria:

* No informed consent,
* Intolerance with respect to ziprasidone or risperidone,
* Contraindications with respect to these substances,
* Gravidity or missing anticonceptive safety
* Substance dependance (excluded nicotin)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2003-11; Study Completion 2006-09

PRIMARY OUTCOMES:
PANSS, SANS, HAMD, GAF, CGI, QTc

SECONDARY OUTCOMES:
Body weight, EPMS, Akathisia,Prolactin, blood pressure, heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Zink, MD, Principal Investigator — Central Institute of Mental Health, Department of Psychiatry, Mannheim, Germany
Locations (1):
- Central Institute of Mental Health, Department of Psychiatry,, Mannheim, Baden-Wurttemberg, Germany